CLINICAL TRIAL: NCT04837378
Title: Effects of Abdominal Massage and In-Bed Exercise on Gastrointestinal Complications and Patient Comfort in Intensive Care Patients Eating Enterally
Brief Title: The Effect of Abdominal Massage and In-bed Exercise on Enteral Nutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Zeliha CENGİZ, Principal Investigator, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021/1839
Record Dates: First submitted 2021-04-02; First posted 2021-04-08 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Patient Engagement
Keywords: Abdominal Massage; Enteral Nutrition; Comfort; In-Bed Exercise; Intensive Care
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Intervention Model Description: In the study, patients will be stratified according to their gender (male and female) status and the blocking process will be performed. 46 patients will be included in each group by repeating the layers formed according to the specified variables 3 times. The stratified patients will be assigned to the experimental and control groups, and the research groups will be written on papers for the determined sets and a lot will be drawn.
  Group 1: Abdominal Massage 2. Group: In-bed Exercise 3. Group: Control
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Abdominal Massage Group (Experimental): Abdominal massage process stage; After the preliminary test data were obtained, the hands were warmed and creamed with vaseline, abdominal massage was applied to the patient in the supine position for 15 minutes. After 24 hours, gastrointestinal complications and comfort parameters were recorded.
  Interventions: Other: Abdominal Massage
- In-bed Exercise Group (Experimental): In-bed exercise process phase; After the pre-test data were obtained, the patient was applied passive in-bed exercises for approximately 15 minutes in all extremities in the supine position. After 24 hours, gastrointestinal complications and comfort parameters were recorded.
  Interventions: Other: In-bed Exercise
- Control Group (No Intervention): Control group stage; Gastrointestinal complications and comfort parameters were recorded in this group at the same time as the experimental groups without any intervention.

INTERVENTIONS:
Other: Abdominal Massage — The massage starts from the left lower quadrant of the sigmoid colon. After the initial tension is removed, deep effloration, petrization and vibration maneuvers are started. Finally, the process is completed in about 15 minutes to cover the entire column.
  Arms: Abdominal Massage Group
Other: In-bed Exercise — In-bed exercises are passive exercises performed by caregivers when the patient is dependent on the bed, that is, when he cannot actively move on his own. These are movements applied to all joints of the upper and lower extremities and in all directions. Exercises are done in all directions on finger joints of both hands, wrists, elbow and shoulder joints, finger joints of both feet, ankles, knee and hip joints.
  Arms: In-bed Exercise Group

SUMMARY:
Enteral nutrition is often preferred in intensive care units, but it brings some potential complications in addition to its benefits. It is stated that abdominal massage and in-bed exercise in intensive care patients can reduce complications related to the gastrointestinal system when performed under appropriate conditions. Considering the ease of application, low cost and non-invasive nature of abdominal massage and in-bed exercises, it is predicted that patients will benefit in case of gastrointestinal complications and positive effects on comfort. It is also thought that these interventions that support independent nursing roles will contribute to the establishment of standards of care and the professionalization process by using evidence-based practices.

This study is conducted to evaluate the effects of abdominal massage and in-bed exercise on gastrointestinal complications and patient comfort in intensive care patients who are fed enterally.

DETAILED DESCRIPTION:
Enteral nutrition is often preferred in intensive care units, but it brings some potential complications in addition to its benefits. It is stated that abdominal massage and in-bed exercise in intensive care patients can reduce complications related to the gastrointestinal system when performed under appropriate conditions. Considering the ease of application, low cost and non-invasive nature of abdominal massage and in-bed exercises, it is predicted that patients will benefit in case of gastrointestinal complications and positive effects on comfort. It is also thought that these interventions that support independent nursing roles will contribute to the establishment of standards of care and the professionalization process by using evidence-based practices.

This study is conducted to evaluate the effects of abdominal massage and in-bed exercise on gastrointestinal complications and patient comfort in intensive care patients who are fed enterally.

The research is planned to be completed between April 15, 2021 and July 15, 2022. The universe of the study, which was conducted as a randomized controlled study model, consisted of patients with intubated enteral nutrition in the internal intensive care units of Diyarbakır Gazi Yaşargil Training and Research Hospital and Dicle University Medical Faculty. Participants were planned to be assigned to the experimental and control groups by stratification and block randomization (Abdominal massage group = 46 participant, in-bed exercise group = 46 participant and control group = 46 participant). Demographic Characteristics Form, Enteral Nutrition Follow-up Form, Richmond Agitation-Sedation Scale, Intensive Care Pain Observation Scale and Comfort Behavior Checklist were used to collect data. According to the characteristics of the data, t test, ANOVA test, Mann Whitney U test and correlation were measured in independent groups.

ELIGIBILITY:
Inclusion Criteria:

* • Patients connected to a mechanical ventilator

  * Patients who started enteral feeding with a nasogastric tube at least 24 hours ago
  * Patients with no injuries to the extremity and abdominal area
  * Patients without intestinal obstruction
  * Patients who have not received abdominal radiotherapy and have not undergone abdominal surgery during the last six weeks
  * Patients with Glasgow Coma Score (GCS) > 3
  * Patients with Acute Physiology and Chronic Health Evaluation (APACHE II)> 16
  * Patients given consent by their first-degree relative

Exclusion Criteria:

* • Patients whose enteral feeding was discontinued during the study

  * Patients who show signs of infection due to VAP or other infections during or before the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
The effect of abdominal massage on gastrointestinal complications | About 6 months
  Abdominal massage was repeated for 3 days, and gastric residual volume, defecation frequency, vomiting number, abdominal distension, constipation and diarrhea status and blood glucose measurement were recorded before each abdominal massage.
The effect of abdominal massage on patient comfort | About 6 months
  Comfort behavior checklist (CBC) consists of 30 behavioral indicators, pain and comfort scores. Minimum score is 25, maximum score is 100. High scores indicate a high level of comfort. Scoring was done before and after abdominal massage.
Effects of in-bed exercise on gastrointestinal complications | About 6 months
  The in-bed exercise was repeated for 3 days and the gastric residual volume, defecation frequency, vomiting number, abdominal distension, constipation and diarrhea status, and blood glucose measurement were recorded in the enteral nutrition follow-up form before each exercise.
The effect of in-bed exercise on patient comfort | About 6 months
  The comfort behavior checklist (CBC) consists of 30 behavioral indicators, pain and comfort scores. Minimum score is 25, maximum score is 100. High scores indicate a high level of comfort. Scoring was done before and after the in-bed exercise.

CONTACTS AND LOCATIONS:
Locations (1):
- SBÜ Gazi Yaşargil Training and Research Hospital, Diyarbakır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This research is a doctoral thesis study. The research is expected to be completed.